CLINICAL TRIAL: NCT04506411
Title: Placebo Controlled Randomized Clinical Trial to Evaluate Efficacy of Turmipure Gold® to Improve Joint Function in Subjects With Distinct Kellgren-Lawrence Knee Radiographic Scores
Brief Title: Turmeric Efficacy for Mobility and Joint Function
Acronym: T-MOTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Givaudan France Naturals (Industry)
Collaborators: Artialis (Industry); Vizera d.o.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0120-118/2020/9
Record Dates: First submitted 2020-07-29; First posted 2020-08-10 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Knee Discomfort; Joint Pain
Keywords: Mobility; Joint function; Turmeric; Curcuminoids
MeSH Terms: conditions — Arthralgia | interventions — Diarylheptanoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TPG (Experimental): 59 participants who meet the eligibility criteria will be randomized under experimental arm and will receive Turmipure GOLD® product during 12 weeks
  Interventions: Dietary Supplement: Turmipure GOLD®
- STE (Active Comparator): 59 participants who meet the eligibility criteria will be randomized under experimental arm and will receive standard turmeric extract 95% curcuminoids (STE) product during 12 weeks
  Interventions: Dietary Supplement: Turmeric rhizome PE 95% curcuminoids
- Control (Placebo Comparator): 59 participants who meet the eligibility criteria will be randomized under experimental arm and will receive placebo (maltodextrin) product during 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Turmipure GOLD® — TPG: Turmipure GOLD® capsules - 4 capsules once daily- as prescribed
  Arms: TPG
Dietary Supplement: Turmeric rhizome PE 95% curcuminoids — STE: Turmeric rhizome PE 95% curcuminoids - 4 capsules once daily- as prescribed
  Arms: STE
Dietary Supplement: Placebo — Placebo: Maltodextrin - 4 capsules once daily- as prescribed
  Arms: Control

SUMMARY:
The objective of the study is to test the capacity of a 12-weeks Turmipure GOLD® supplementation to reduce joint discomfort.

DETAILED DESCRIPTION:
The aim of this clinical study is to determine whether oral administration of Turmipure GOLD® can contribute to the improvement of mobility and joint function in adult population with knee discomfort and with distinct Kellgren-Lawrence (K&L) knee radiographic scores.

ELIGIBILITY:
Inclusion Criteria:

* Consent to the study and to comply with study product
* Who have a BMI between 18 and 32 kg/m²
* Who has mild to moderate knee pain for at least 3 months before enrollment (VAS between 40 to 70 on 100mm scale after respecting a washout period depending on the half-life of the excluded medications)
* Who has radiographic evidence of Kellgren-Lawrence score 0, 1, 2 and 3 in the tibio-femoral compartment of the target knee
* Who is able to perform the physical performance-based tests and understands all questions from the WOMAC questionnaire
* Who is willing to refrain from taking any pain reliever (OTC or prescription) and other pharmacological, nutritional agent (e.g. glucosamine), device or therapy (e.g. acupuncture) which may influence the study outcome during the entire trial (other than determined authorized rescue medication)
* Who is willing to not change dietary habits, level of physical activity (including any heavy physical work with high loading of the knee joints) and body weight

Exclusion Criteria:

* Subjects with any clinically significant levels of the safety parameters at screening
* Pregnant or lactating females, or wishing to become pregnant during the study
* Subject with joint pain related to some predisposing conditions that have adversely altered the joint tissues often due to a specific cause
* Subject with Kellgren-Lawrence grade 4 in the tibio-femoral compartment of the target knee
* Who has clinically apparent tense effusion of the target knee or other joint
* Who has/had viscosupplementation in any joint including the target knee or other joint within 6 months prior to screening
* Who has concomitant inflammatory disease or other condition that affects the joints deemed exclusionary by the Principal Investigator (e.g. rheumatoid arthritis, metabolic bone disease, psoriasis, gout, symptomatic chondrocalcinosis and active infection, etc…)
* Who has symptomatic osteoarthritis of the contralateral knee that is not responsive to paracetamol and requires other therapy
* Who is taking any treatment/supplementation which may interfere with study conduct and interpretation of study results (4-weeks washout, e.g. glucosamine, chondroitin, corticosteroids) except calcium and vitamin D supplements
* Who is under any medical condition deemed exclusionary by the Principal Investigator
* Subject has a history of drug and / or alcohol abuse at the time of enrollment
* Change of dietary habit within the preceding month
* Subject with known organic disease, including an inflammatory bowel disease, a benign or malign tumor of intestine or colon and significant systemic disease
* Subject currently involved in any other clinical trial or having participated in a trial within the preceding 90 days
* Subject with known allergy to components of the test product
* Subject has any concurrent medical or psychiatric condition that, in the opinion of the Investigator, would compromise his/her ability to comply with the study requirements
* History of cancer within the last 5 years, except basal cell carcinoma, non-squamous skin carcinoma, prostate cancer or carcinoma in situ with no significant progression over the past 2 years
* Significant cardiovascular, pulmonary, renal, liver, infectious disease, immune disorder, or metabolic/endocrine disorders or other disease that would preclude supplement ingestion and/or assessment of safety and the study objectives
* Current illnesses which could interfere with the study (e.g. prolonged severe diarrhea, regurgitation/severe, difficulty swallowing)
* Who is taking any anticoagulant or heparin treatment

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Change in WOMAC™ Pain | 12-weeks
  Knee joint pain discomfort assessed with the validated Western Ontario and McMaster University questionnaire (WOMAC) using its visual analogue scale version (VAS). The WOMAC VA 3.1 Pain subscore (WOMAC A) ranges from 0 to 100 mm (averaging five VAS 0-100 mm) with higher scores indicating more pain.

SECONDARY OUTCOMES:
Change in WOMAC™ Stiffness | 12-weeks
  Knee joint stiffness assessed with the validated Western Ontario and McMaster University questionnaire (WOMAC) using its visual analogue scale version (VAS). The WOMAC VA 3.1 Stiffness subscore (WOMAC B) ranges from 0 to 100 mm (averaging two VAS 0-100 mm) with higher scores indicating more stiffness.
Change in WOMAC™ Physical function | 12-weeks
  Knee joint physical function assessed with the validated Western Ontario and McMaster University questionnaire (WOMAC) using its visual analogue scale version (VAS). The WOMAC VA 3.1 Physical function subscore (WOMAC C) ranges from 0 to 100 mm (averaging seventeen VAS 0-100 mm) with higher scores indicating more stiffness.
Change in WOMAC™ Global Index | 12-weeks
  Knee joint global discomfort assessed through the sum of WOMAC A (pain), WOMAC B (stiffness) and WOMAC C (physical function) subscores. The WOMAC Global Index score ranges from 0 to 2400 mm (summing up twenty-four VAS 0-100 mm), with higher scores indicating higher disease burden.
Pain intensity at rest | 12-weeks
  The pain intensity at rest is assessed using a VAS ranging from 0 to 100 mm, with higher scores indicating more pain.
Pain intensity while walking | 12-weeks
  The pain intensity while walking is assessed using a VAS ranging from 0 to 100 mm, with higher scores indicating more pain.
"Patient Global Assessment" (PGA) | 12-weeks
  The "Patient Global Assessment" (PGA) is the global assessment on joint discomfort and is assessed using a VAS ranging from 0 to 100 mm, with higher scores indicating more pain.
OMERACT-OARSI criteria | 12-weeks
  Evaluation of the response to supplementation
30s Chair Stand Physical Performance | 12-weeks
  Evaluation of the maximum number of chair stand repetitions possible in a 30 second period. Scoring results in a wide range of skill levels from 0, for those who cannot complete a single repetition and values greater than 20 for the well prepared individuals.
40m Fast-paced Walked Physical Performance | 12-weeks
  A fast-paced walking test that is timed over 4 x 10m (33 ft) for a total 40 m (132 ft) evaluating the ability to walk quickly over short distances. Time of one test trial is recorded and expressed as speed m/s by dividing distance (40m) by time (s).
Stair Climb Physical Performance | 12-weeks
  Evaluates the time (in seconds) it takes to ascend and descend a flight of stairs. Timing begins on the signal to start and terminates when the participant returns with both feet to the ground level and the total time to ascend and descend steps for 1 test trial is recorded to nearest 100th of a second.
Time up & Go Physical Performance | 12-weeks
  Evaluates the time (seconds) taken to rise from a chair, walk 3 m (9 ft 10 inches), turn, walk back to the chair, then sit down. Timing starts on the signal to start and terminates once the participant sits back down fully with their back resting on the back of the chair. Two trials are performed and the faster of the 2 trials is recorded to nearest 10th of a second.
Quality of Life evaluation | 12-weeks
  Evaluation of Quality of life through SF-36 (RAND version), which is a set of generic, coherent, and easily administered quality-of-life measures. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability and the higher the score the less disability.
Clinical Global Impression of Change (CGIC) | 12-weeks
  Physician assessment of joint swelling and range of motion (ROM) for knee extension/flexion, indicating the perceived change over the treatment period. The clinician is requested to choose one of seven categories. Scores range from very much improved to very much worse.
Assessment of use of rescue medicine | 12-weeks
  Evaluation of associated treatments needed to manage joint complains

CONTACTS AND LOCATIONS:
Overall Officials: Matija Tomšič, Prof., MD, Study Chair — Univerzitetni klinični center Ljubljana, Klinični oddelek za revmatologijo, Ljubljana, Slovenia; Samo K Fokter, MD, Principal Investigator — Univerzitetni klinični center Maribor, Oddelek za ortopedijo
Locations (8):
- Croatia (2):
  - Poliklinika Aviva, Zagreb
  - Poliklinika Idassa, Zagreb
- Slovenia (6):
  - Ortopedska bolnišnica Valdoltra, Ankaran
  - Splošna bolnišnica Jesenice, Oddelek za ortopedijo, Jesenice
  - Bisturmed, d.o.o., Ortopedija in fizioterapija, Koper
  - Poliklinika Nobilis, d.o.o., enota LJ, Ortopedska ambulanta, Ljubljana
  - Medicinsko termalni center Fontana, d.o.o., Ortopedska ambulanta, Maribor
  - Univerzitetni klinični center Maribor, Oddelek za ortopedijo, Maribor

IPD SHARING:
Plan to Share IPD: Undecided
To revisit after investigation period